CLINICAL TRIAL: NCT06787365
Title: Questionnaire for the Assessment of Risk Factors Associated with Endometriosis in Adolescent Women Diagnosed with Endometriosis
Brief Title: Questionnaire for the Assessment of Risk Factors Associated with Endometriosis in Adolescent Women with Endometriosis
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: QuestionENDO
Record Dates: First submitted 2024-12-03; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Endometriosis
Keywords: Endometriosis; Gynaecology; Questionnaire; Risk factors; Painful symptoms
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Patients with endometriosis
- Control group: Patients without endometriosis

SUMMARY:
A number of risk factors that may be associated with endometriosis in adolescents (medical history and symptoms) are reported in the literature, but no overall estimate of disease risk has been developed.

Providing a tool for assessing risk factors associated with endometriosis in adolescents by estimating disease risk could aid the clinician in diagnosis and reduce diagnostic delay

DETAILED DESCRIPTION:
Although more than 60% of adult women with endometriosis report that their painful symptoms appeared before the age of 20, early diagnosis, particularly in adolescent girls, is still a challenge for doctors. The reasons for this delay include inadequate knowledge of the disease among healthcare professionals, the social and health normalisation of menstrual pain, and the peculiar aspects of the disease in adolescent patients. The adolescent patient with endometriosis presents particular anamnestic, familial and personal risk factors, as well as peculiar symptoms such as non-specific abdominal pain, acyclic pelvic pain, gastrointestinal symptoms, migraine, in addition to those classically reported in adulthood.

It may therefore be useful to identify a predictive model of the onset of endometriosis based on the risk factors currently recognised in the literature (anamnestic data) and on the results of a questionnaire to be submitted to adult women (aged between 20 and 50 years), with endometriosis (group 1) and without a diagnosis of endometriosis (group 2), concerning symptoms experienced in adolescence

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age between 20 and 50 years
* Clinical and ultrasound diagnosis of endometriosis for the study group and exclusion of endometriosis for the control group (examination and ultrasound performed according to the IDEA study criteria)
* Acquisition of informed consent for participation in the study and processing of personal data

Exclusion Criteria:

- Women suffering from other conditions responsible for pelvic pain (uterine fibromatosis, current or previous pelvic inflammatory disease, ovarian cysts of a non-endometriotic nature, irritable bowel syndrome, inflammatory bowel disease, interstitial cystitis)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with and without a diagnosis of endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Predictive model of endometriosis onset risk | During the first visit after enrollment
  Predictive model of the occurrence of endometriosis based on the risk factors currently recognised in the literature (anamnestic data) and the results of a questionnaire consists of 28 multiple-choice questions, concerning symptoms experienced in adolescence

CONTACTS AND LOCATIONS:
Overall Officials: Simona Del Forno, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Senese, Siena, Siena